CLINICAL TRIAL: NCT07135336
Title: Incidence of Postoperative Cognitive Decline in Surgical Patients With Preexisting Cognitive Impairment: A Prospective Cohort Study
Brief Title: Incidence of Postoperative Cognitive Decline in Patients With Preexisting Cognitive Impairment
Status: Recruiting | Type: Observational
Sponsor: Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025（134）
Record Dates: First submitted 2025-06-25; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Cognitive and Behavioral Impairment
Keywords: postoperative cognitive decline; preexisting cognitive impairment
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preexisting Cognitive Impairment (PreCI) Group: Patients aged 60 years and older with preexisting cognitive impairment undergoing elective non-cardiac surgery under general anesthesia. These patients will receive standard perioperative care without any additional intervention. Cognitive function and neuropsychiatric status will be assessed before surgery, and at 3 and 12 months after surgery to determine the incidence of postoperative cognitive decline (POCD).
  Interventions: Procedure: surgery
- Normative Population: Cognitively normal individuals recruited from inpatients and outpatients of Peking University Shenzhen Hospital. These participants will not undergo surgery but will complete the same cognitive assessments at baseline, 3 months, and 12 months. The normative data will be used to calculate the Reliable Change Index (RCI) for identifying clinically significant cognitive decline in the PreCI group.
  Interventions: Other: norma

INTERVENTIONS:
Procedure: surgery — Patients with preexisting cognitive impairment undergoing elective non-cardiac surgery under general anesthesia.
  Groups: Preexisting Cognitive Impairment (PreCI) Group
Other: norma — Cognitively normal individuals who do not undergo surgery but complete the same cognitive assessments at baseline, 3 months, and 12 months for normative reference.
  Groups: Normative Population

SUMMARY:
This study aims to find out how often memory and thinking problems happen after surgery in people who already have memory issues before their operation. These memory problems are called postoperative cognitive decline (POCD). Older adults with memory problems before surgery may be more likely to have trouble with thinking, memory, and daily activities after their operation. This study will follow patients who already have memory problems before surgery and see how their thinking and memory change after surgery. The results will help doctors better understand how to care for these patients before, during, and after surgery.

DETAILED DESCRIPTION:
This is a single-center, prospective, single-arm cohort study designed to estimate the incidence of postoperative cognitive decline (POCD) in patients aged 60 years and older with preexisting cognitive impairment undergoing elective non-cardiac surgery under general anesthesia.

To calculate the incidence of POCD, a normative population of cognitively normal individuals will be recruited to provide reference data for the expected range of cognitive change over time in the absence of surgery. This normative sample is not a control group for intervention comparison but is used to establish population-based norms for cognitive test score changes.

Study Procedures:

Preoperative assessment (1 day before surgery):

Patients will be screened using the Mini-Cog test. Those with scores ≤1 will be further evaluated with the Mini-Mental State Examination (MMSE) and Beijing version of the Montreal Cognitive Assessment (MoCA-B).（This threshold is based on the Chinese expert consensus scoring criteria, which differ slightly from the international standard. According to the Chinese algorithm, a score of ≤1 encompasses cases where the clock drawing is incorrect and one to two words are recalled, or when no words are recalled at all, aligning functionally with a score of ≤2 in the international system. Therefore, our inclusion criterion of ≤1 under the Chinese system is equivalent in diagnostic implication to the widely accepted international cutoff of ≤2, which indicates high likelihood of cognitive impairment.) Eligible participants will be enrolled after informed consent is obtained. Neuropsychiatric symptoms will be assessed using the Neuropsychiatric Inventory-Questionnaire (NPI-Q). Dementia severity and functional ability will be evaluated using the Clinical Dementia Rating (CDR), Basic Activities of Daily Living (BADL), and Instrumental Activities of Daily Living (IADL) scales.

Intraoperative data collection:

Information regarding surgery and anesthesia will be obtained from the electronic medical records.

Postoperative follow-up (at 3 and 12 months):

All participants will undergo cognitive assessments using the MMSE and MoCA-B. Neuropsychiatric symptoms, dementia severity (if applicable), and functional abilities will also be reassessed. Follow-up will be scheduled to minimize participant burden, and home-based assessments will be arranged when necessary. Remote assessments will be documented if used.

Normative Population:

Cognitively normal individuals will be recruited from inpatients and outpatients of Peking University Shenzhen Hospital. They will undergo cognitive assessments at baseline, 3 months, and 12 months to provide normative data for the calculation of standardized cognitive changes.

Primary Outcome:

The primary outcome is the incidence of POCD at 3 months after surgery. Following the nomenclature recommendations by Evered et al., POCD is defined as objectively measurable cognitive decline occurring between 3 months and 7.5 years after surgery. The diagnosis of POCD in this study will be based on the Reliable Change Index (RCI), a standardized statistical method that accounts for normal variability and practice effects over time.

RCI is calculated as:

RCI = (ΔX_patient - Δμ_normative) / σ_normative

Where ΔX_patient is the individual's change score, Δμ_normative is the mean change in the normative group, and σ_normative is the standard deviation of change scores in the normative group.

A patient will be considered to have POCD if either:

At least two cognitive domains show an RCI ≤ -1.96, or

The combined Z-score of all cognitive tests is ≤ -1.96.

Follow-up Management and Missing Data Handling:

Participants will be followed at 3 and 12 months. If a participant is unable to attend, alternative arrangements will be made. Loss to follow-up will be documented with reasons, and missing data will be addressed using sensitivity analyses.

ELIGIBILITY:
1. Preexisting Cognitive Impairment (PreCI) Surgical Group

   Inclusion Criteria:
   * Age ≥ 60 years
   * Preoperative screening with MMSE and MoCA-B indicating mild cognitive impairment (MCI) or mild dementia
   * Undergoing elective non-cardiac surgery under general anesthesia

   Exclusion Criteria:
   * Expected difficulty in completing neuropsychological assessments (e.g., inability to communicate in Mandarin, blindness, or deafness)
   * Usual residence outside Shenzhen
2. Normative Reference Group

Inclusion Criteria:

* Age ≥ 60 years
* No history of general anesthesia surgery within the past 12 months
* Mini-Cog score > 1

Exclusion Criteria:

* Planned elective surgery under general anesthesia within the next 12 months
* History of suspected or diagnosed cognitive impairment, or screening indicating cognitive impairment using MMSE and MoCA-B
* Expected difficulty in completing neuropsychological assessments (e.g., inability to communicate in Mandarin, blindness, or deafness)
* Usual residence outside Shenzhen

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 60 years and older with preexisting cognitive impairment undergoing elective non-cardiac surgery under general anesthesia at Peking University Shenzhen Hospital will be recruited between June 2025 and December 2027. A normative reference group of cognitively normal elderly individuals, matched by age and sex, will also be enrolled from the same hospital during the same period. All participants must reside in Shenzhen and be able to communicate in Mandarin.
Sampling Method: Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Cognitive Decline (POCD) at 3 Months | 3 months after surgery
  The primary outcome is the incidence of objectively measurable postoperative cognitive decline (POCD) at 3 months in patients with preexisting cognitive impairment undergoing elective non-cardiac surgery under general anesthesia. The diagnosis of POCD will follow the nomenclature recommendations by Evered et al., which define POCD as cognitive decline occurring between 3 months and 7.5 years after surgery, determined by standardized score changes compared with a normative reference population.
  In this study, POCD will be identified using the Reliable Change Index (RCI), calculated as:
  RCI = (ΔX_patient - Δμ_normative) / σ_normative
  A patient will be diagnosed with POCD if:
  At least two cognitive domains show an RCI ≤ -1.96, or
  The combined Z-score of all cognitive tests is ≤ -1.96.

SECONDARY OUTCOMES:
Incidence of POCD at 12 Months | 12 months after surgery
  Incidence of objectively measurable POCD at 12 months postoperatively, assessed using the same criteria as the primary outcome (RCI method).
Neuropsychiatric Symptoms Assessed by NPI-Q | 3 and 12 months after surgery
  Neuropsychiatric symptoms will be evaluated using the Neuropsychiatric Inventory-Questionnaire (NPI-Q), based on caregiver or informant reports. It assesses the presence, severity, and caregiver distress associated with 12 neuropsychiatric symptoms commonly seen in patients with cognitive impairment. For each symptom, severity is rated on a scale from 1 to 3 (1 = mild, 2 = moderate, 3 = severe), with a total severity score ranging from 0 to 36. Higher scores indicate more severe neuropsychiatric symptoms.
Functional Ability Assessed by The Barthel Index | 3 and 12 months after surgery
  The Barthel Index (BI) in an informant report was used for measuring basic ADL actual performance in this study. The BI is a questionnaire that consists of ten items: feeding, bathing, grooming, dressing, bowels, bladder, toilet use, transfer, mobility, and stairs. The summary score ranges from 0 to 100, with lower scores indicating a poorer basic ADL performance
Dementia Severity Assessed by CDR | 3 and 12 months after surgery
  The Clinical Dementia Rating (CDR) will be used to assess the severity of dementia by evaluating six cognitive and functional domains. Scores range from 0 (no impairment) to 3 (severe dementia). CDR scores will be recorded at each follow-up.
Instrumental activities of daily living by The Lawton IADL | 3 and 12 months after surgery
  Instrumental activities of daily living (IADL) will be assessed using the Lawton-Brody Instrumental Activities of Daily Living Scale, a widely validated and reliable tool for evaluating functional independence in older adults. The scale includes eight domains: using the telephone, shopping, preparing meals, housekeeping, laundry, using transportation, managing medications, and handling finances. The assessment will be conducted through informant-based interviews or direct patient self-report, depending on cognitive status. Each item is scored dichotomously (0 or 1): 1 point indicates independence in performing the activity 0 points indicates dependence or inability to perform the activity. The total score ranges from 0 to 8, with higher scores indicating greater functional independence. A total score ≤6 may suggest moderate to severe functional impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data may be considered for sharing upon reasonable request after the study results have been published, subject to additional ethical approval.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT07135336/Prot_SAP_000.pdf